CLINICAL TRIAL: NCT01703949
Title: A Pilot Study of Weekly Brentuximab Vedotin or Brentuximab Vedotin Plus Nivolumab Every 3 Weeks in Patients With CD30+ Malignancies Refractory to Every ≥ 3 Week Brentuximab Vedotin
Brief Title: Brentuximab Vedotin With or Without Nivolumab in Treating Patients With Relapsed or Refractory CD30+ Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7808; NCI-2012-01696 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 7808 (Other: Fred Hutch/University of Washington Cancer Consortium); RG1713010 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2012-10-08; First posted 2012-10-11 (Estimated); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Recurrent Hodgkin Lymphoma; Recurrent Non-Hodgkin Lymphoma; Refractory Hodgkin Lymphoma; Refractory Non-Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin | interventions — Brentuximab Vedotin; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (brentuximab vedotin) (Experimental): Patients receive brentuximab vedotin IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Brentuximab Vedotin; Other: Laboratory Biomarker Analysis
- Arm B (brentuximab vedotin, nivolumab) (Experimental): Patients receive brentuximab vedotin IV over 30 minutes and nivolumab IV over 30-60 minutes on day 1. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Brentuximab Vedotin; Other: Laboratory Biomarker Analysis; Biological: Nivolumab

INTERVENTIONS:
Drug: Brentuximab Vedotin — Given IV
  Other Names: ADC SGN-35; Adcetris; Anti-CD30 Antibody-Drug Conjugate SGN-35; Anti-CD30 Monoclonal Antibody-MMAE SGN-35; Anti-CD30 Monoclonal Antibody-Monomethylauristatin E SGN-35; cAC10-vcMMAE; SGN-35
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo; CMAB819; Nivolumab Biosimilar CMAB819
  Arms: Arm B (brentuximab vedotin, nivolumab)

SUMMARY:
This phase II pilot trial studies how well brentuximab vedotin with or without nivolumab works in treating patients with CD30+ lymphoma that has come back after a period of improvement or does not respond to treatment. Biological therapies, such as brentuximab vedotin, may stimulate the immune system in different ways and stop cancer cells from growing. Monoclonal antibodies, such as nivolumab may interfere with the ability of tumor cells to grow and spread. Giving brentuximab vedotin with or without nivolumab may work better in treating patients with CD30+ lymphoma.

DETAILED DESCRIPTION:
OUTLINE:

ARM A (CLOSED TO ACCRUAL): Patients receive brentuximab vedotin intravenously (IV) over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive brentuximab vedotin IV over 30 minutes and nivolumab IV over 30-60 minutes on day 1. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 3-5 weeks, every 3 months for 1 year, and then every 6 months for 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory CD30+ lymphoma that has either achieved < PR to brentuximab vedotin (minimum of 2 cycles), progressed while receiving brentuximab vedotin, or progressed within 6 months of the last dose of brentuximab vedotin
* Documented expression of CD30 on tumor cells
* Absolute neutrophil count (ANC) > 1,000/uL
* Platelets > 50,000/uL
* Serum creatinine < 1.5 mg/dL OR creatinine clearance > 60 mL/min
* Bilirubin < 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 x ULN
* Measurable disease by computed tomography (CT) or similar (e.g. magnetic resonance imaging [MRI]) criteria (> 1.5 cm). (Patients with cutaneous lymphoma only require measurable disease by Olsen Criteria)
* Age >= 18 yrs at the time of the first dose of study drug
* Resolution of all non-hematologic brentuximab vedotin-related and nivolumab-related adverse events (AEs) to < Grade 2
* All patients must be informed of the investigational nature of this study and have given written consent in accordance with institutional and federal guidelines
* Patients must be anticipated to complete at least 2 cycles of chemotherapy on study
* Expected survival if untreated of > 90 days

Exclusion Criteria:

* Prior transplant within 100 days
* Radioimmunotherapy within 12 weeks
* Known human immunodeficiency virus (HIV) or hepatitis B positivity or prior progressive multifocal leukoencephalopathy (PML)
* Active infection or other medical condition which would preclude treatment in the opinion of the principal investigator; this would include a corrected diffusing capacity of the lungs for carbon monoxide (DLCO) of < 60% predicted or symptomatic interstitial lung disease
* Eastern Cooperative Oncology Group (ECOG) performance status > 2
* Known active central nervous system (CNS) involvement
* Peripheral neuropathy > grade 1 if due to brentuximab vedotin or any peripheral neuropathy > grade 2
* Intolerance to brentuximab vedotin
* Concurrent use of other anti-cancer agents or experimental treatments
* No current or prior autoimmune disease with the exception of vitiligo and autoimmune alopecia (Arm B only)
* Pregnancy or breastfeeding; (females of childbearing potential must have a negative serum or urine beta human chorionic gonadotropin [beta-hCG] pregnancy test result within 7 days prior to the first dose of brentuximab vedotin; females with false positive results and documented verification that the patient is not pregnant are eligible for participation; females of non-childbearing potential are those who are postmenopausal greater than 1 year or who have had a bilateral tubal ligation or hysterectomy; females of childbearing potential and males who have partners of childbearing potential must agree to use 2 effective contraceptive methods during the study and for 6 months following the last dose of brentuximab vedotin or 6 months following the last dose of nivolumab, whichever is later)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-03-20 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2030-06-03 (Estimated)

PRIMARY OUTCOMES:
Overall response rate as measured by the Cheson 2007 criteria | For Arm A: Up to 5 weeks after completion of study treatment. For Arm B: within 6 months following treatment.
  No formal statistical measures will be pre-specified. This protocol will be deemed a "success" if the absolute response rate in this group of patients is ≥20% in Arm A or ≥40% in Arm B.

CONTACTS AND LOCATIONS:
Overall Officials: Ajay K. Gopal, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States